CLINICAL TRIAL: NCT00194454
Title: Psychosocial/Behavioral Intervention in PSD
Brief Title: Psychosocial/Behavioral Intervention in Post-Stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Pamela H. Mitchell, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00-3203-V 06; 5R01NR007755-04 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Stroke
Keywords: Depressive symptoms; Behavior and behavior mechanisms; Recovery
MeSH Terms: conditions — Stroke; Depression; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nine session psychosocial/behavioral counseling with homework
  Interventions: Behavioral: Modified cognitive behavioral therapy plus problem-solving
- 2 (Active Comparator): Usual clinic care with booklet describing depression following stroke
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: Modified cognitive behavioral therapy plus problem-solving — 9 sessions with a psychosocial nurse practitioner in which participants learn to use behavioral strategies and specific problem-solving approaches to reduce or prevent behavioral and mood disturbances characteristic of stroke.
  Arms: 1
Other: usual care — Usual care with primary provider plus a booklet about mood and behavioral changes following stroke
  Arms: 2

SUMMARY:
The primary aim of this study is to determine the effect of a nurse-delivered psychosocial/behavioral intervention on reduction of depression in community dwelling post-stroke patients. We expect the combined behavioral and pharmacologic intervention to be more effective than pharmacotherapy alone in sustaining the improvement in depression for the experimental group. Secondary aims are to examine the effect of the psychosocial/behavioral intervention time course and sustainability of response to treatment, effect on limitations in ability, limitation in participation and overall stroke impact in community-dwelling post-stroke patients, and to compare ischemic stroke survivors who are and are not depressed within the first four months following stroke by their 5-HTTLPR genotypes (s/s, s/l, or l/l).

DETAILED DESCRIPTION:
150 patients at University of Washington affiliated hospitals who are found to be depressed by DSMIV criteria within the first four months following ischemic stroke will be invited to join the study, and randomly assigned to a problem-solving/pleasant events intervention provided by an advanced practice nurse, or to regular clinic follow-up. Both groups will receive standard antidepressant treatment and written materials from the American Stroke Association, and will be assessed for up to two years following the study. The primary outcome is reduction in depression at 12 months following stroke. Secondary outcomes are reductions in limitations in activity (Barthel Index), reduction in limitation in participation (Stroke Impact Scale) and overall stroke impact (Stroke Impact Scale) at 6, 12, and 24 months post- stroke. We hypothesize that all patients will improve their mood and functional ability related to their post-stroke standard treatment, but that those who receive the psychosocial intervention will have significantly greater improvement in mood, functional ability, social participation, and less overall stroke impact at all follow-up measurement. A supplemental aim is to expand aim 4 of the parent study, adding SERT genotype to our list of factors that might influence treatment outcome for PSD. Further, since we are screening both depressed and not depressed stroke survivors for this study, we will add a fifth aim: to compare ischemic stroke survivors who are and are not depressed within the first four months following stroke by their 5-HTTLPR genotypes (s/s, s/l, or l/l).

ELIGIBILITY:
Inclusion Criteria:

Ischemic stroke within previous 4 months Screens positive for depressive symptoms by Geriatric Depression Scale Able to provide informed consent -

Exclusion Criteria:

Subarachnoid or intracranial hemorrhagic stroke Global aphasia Reduced level of consciousness (GCS <15)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2002-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Reduction in depression (Hamilton Depression Rating Scale)at 12 months following stroke. | 12 months following stroke

SECONDARY OUTCOMES:
Reduction in limitations in activity (Barthel Index)6, 12, 24 months | 6, 12, 24 months following intervention
Reduction in limitation in participation (Stroke Impact Scale)6, 12, 24 months | 6, 12, 24 months following intervention
Overall stroke impact (Stroke Impact Scale)6,12,24 months post- stroke. | 6, 12, 24 months following stroke

CONTACTS AND LOCATIONS:
Overall Officials: Pamela H Mitchell, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Mitchell PH, Teri L, Veith R, Buzaitis A, Tirschwell D, Becker K, Fruin M, Kohen R, Cain KC. Living well with stroke: design and methods for a randomized controlled trial of a psychosocial behavioral intervention for poststroke depression. J Stroke Cerebrovasc Dis. 2008 May-Jun;17(3):109-15. doi: 10.1016/j.jstrokecerebrovasdis.2007.12.002. PMID 18436150
- [Derived] Kohen R, Cain KC, Buzaitis A, Johnson V, Becker KJ, Teri L, Tirschwell DL, Veith RC, Mitchell PH. Response to psychosocial treatment in poststroke depression is associated with serotonin transporter polymorphisms. Stroke. 2011 Jul;42(7):2068-70. doi: 10.1161/strokeaha.110.611434. PMID 21847802
- [Derived] Mitchell PH, Veith RC, Becker KJ, Buzaitis A, Cain KC, Fruin M, Tirschwell D, Teri L. Brief psychosocial-behavioral intervention with antidepressant reduces poststroke depression significantly more than usual care with antidepressant: living well with stroke: randomized, controlled trial. Stroke. 2009 Sep;40(9):3073-8. doi: 10.1161/STROKEAHA.109.549808. Epub 2009 Aug 6. PMID 19661478